CLINICAL TRIAL: NCT05196867
Title: A Randomized, Prospective Study of a Behaviorally-based Tailored Disease Management Intervention vs Control in Patients With Risk Factors for Liver Disease
Brief Title: Liver Cancer Prevention Randomized Control Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Cancer Prevention Research Institute of Texas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2021-1015; NCI-2021-14391 (Other: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-12-29; First posted 2022-01-19 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Liver Diseases; Fibrosis, Liver; Cirrhosis, Liver
MeSH Terms: conditions — Liver Diseases; Liver Cirrhosis | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Immediate Intervention (Experimental): participants will receive the 6 months intervention immediately
  Interventions: Behavioral: Intervention Group
- Arm 2: Delayed Intervention (Experimental): participants will receive the intervention after the 6-month follow-up visit
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: Intervention Group — Participants in the intervention group will receive (1) weekly telephone or videoconference coaching; (2) health education print materials and tip sheets;(3) navigation to programs and resources to help participants meet behavioral goals (e.g., fitness events, classes and webinars, etc); (4) text messages related to behavioral skills; (5) a Fitbit activity tracker and Aria scale; (6) resistance tubes and instructional video for strengthening exercise (if resistance exercise module is chosen); and (7) tools to manage portion sizes.
  Arms: Arm 1: Immediate Intervention
Behavioral: Control Group — Patients in the control arm will initially receive written education material about the risk factors for liver cancer and management options. They will be offered the intervention after they complete the 6-month assessment.
  Arms: Arm 2: Delayed Intervention

SUMMARY:
To determine the effectiveness of a behaviorally-based tailored disease management intervention in patients with fibrosis or steatosis and risk factors for cirrhosis.

DETAILED DESCRIPTION:
Hypothesis: A technology-assisted self-management intervention that addresses diet, physical activity, alcohol use, and medication adherence can produce regression in fibrosis as measured by FIB-4 in patients with fibrosis or steatosis and risk factors for cirrhosis, including chronic hepatitis B virus (HBV) or hepatitis C virus (HCV) infection, alcohol use, or non-alcoholic fatty liver disease (NAFLD).

Primary objective:

To test the effect of the behavioral intervention on fibrosis in a randomized trial. We will randomize eligible HOPE Clinic patients to (i) a 6-month self-management intervention to help participants implement behavioral changes to manage their disease or (ii) a wait-list control group that will receive the intervention after their 6-month assessment.

Secondary objective:

Evaluate changes in behavioral risk factors for liver fibrosis or steatosis (body composition, physical activity, diet, medication adherence, alcohol use), metabolic syndrome, and patient activation and other behavioral determinants.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of steatosis (CAP score ≥ 290 by vibration controlled transient elastography) OR Evidence of liver fibrosis (FIB-4 index ≥ 1.6 or fibrosis grade ≥ F2 by vibration controlled transient elastography [F2 score ≥ 8kPa]) AND meets one of the following criteria: i. overweight or obese (BMI≥23 in Asians or BMI≥25 in other racial groups), OR ii. presence of type II diabetes mellitus, OR iii. lean/normal weight with presence of at least two metabolic risk abnormalities, OR:

1. Waist circumference ≥90/80 cm in Asians or ≥102/88 cm in other racial groups)
2. Blood pressure ≥130/85 mmHg or specific drug treatment
3. Plasma triglycerides ≥150 mg/dl or specific drug treatment
4. Plasma HDL-cholesterol <40 mg/dl for men and <50 mg/dl for women, or specific drug treatment
5. Prediabetes (fasting glucose levels 100-125 mg/dl , or HbA1c 5.7-6.4% ) iv. AUDIT-C ≥4 for men and ≥3 for women AND AUDIT-10 = 8-15

AND/OR 2. Evidence of liver fibrosis (FIB-4 index ≥ 1.6 or fibrosis grade ≥ F2 by vibration controlled transient elastography) and presence of one of the following:

1. chronic HBV (HBsAg+ or taking anti-HBV therapy), or
2. chronic HCV (1. detectable HCV RNA > 4 months or a 2. history of HCV infection and taking anti-HCV therapy)

   3. At least 18 years old 4. Speak and read English or Spanish 5. Access to smartphone with data plan or Wi-Fi access 6. Willing to receive up to 12 text messages per week

   Exclusion Criteria:
   1. Pregnant or planning to become pregnant in next 12 months (by self-report)
   2. Medical contraindications to home-based exercise or low-fat, high-vegetable-and-fruit diet
   3. Recent or planned surgery that would interfere with home-based exercise or a low-fat, high vegetable and fruit diet
   4. Current or prior history of primary liver cancer or cancer that is metastatic to the liver
   5. AUDIT-10 score >15
   6. Family or household member already enrolled into study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in FIB-4 score | up to 6 months
  a serum-based biomarker of fibrosis

CONTACTS AND LOCATIONS:
Overall Officials: Karen Basen-Engquist, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org